CLINICAL TRIAL: NCT02008305
Title: Comparison of Two Protocols of Optimization of X Ray Radiations in Pediatric Interventional Neuroradiology
Acronym: MINIRAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC/DM_MPN_2012-4
Record Dates: First submitted 2013-12-03; First posted 2013-12-11 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Occlusion or Malformation of a Cerebral Vessel
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- protocol of optimization ALARA (Experimental): protocol of optimization ALARA protocol of optimization of doses
  Interventions: Device: protocol of optimization ALARA
- protocol of opimization Philips (Active Comparator): protocol of optimization Philips usual protocol of optimization of doses
  Interventions: Device: protocol of optimization Philips

INTERVENTIONS:
Device: protocol of optimization ALARA
  Arms: protocol of optimization ALARA
Device: protocol of optimization Philips
  Arms: protocol of opimization Philips

SUMMARY:
Interventional Neuroradiology replaces surgery. This technology requires various exposition to X rays : number of X rays photographs, radioscopy, distance between patient and detector, speed of acquisition of X-rays photographs, high tension and intensity.

The manipulator must find the right balance between quality of photographs and dose delivered to the patient (optimization).

Children are particularly exposed to these risks of irradiation (sensitivity to X-rays and long life expectancy with risks. So, it is fundamental to optimize the dose delivered during the procedures.

The investigators propose to analyse a study comparing two protocols of optimization of doses. The investigators' hypothesis is that the protocol experimented in this trial allows less radiation of the children, compared to the usual protocol.

ELIGIBILITY:
Inclusion Criteria:

* malformation or occlusion of a cerebral vessel requiring interventional Neuroradiology

Exclusion Criteria:

* opposition ot the parent(s) to the participation of their child in the trial and/or no social security.

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2013-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the average dose per child, according to the protocol | maximum one day per patient

SECONDARY OUTCOMES:
number of X-rays photographs according to the protocol, quality of photographs according to the protocol, | maximum one day per patient

OTHER OUTCOMES:
number of interrupted dosing | one day per patient

CONTACTS AND LOCATIONS:
Overall Officials: Michel Piotin, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation ophtalmique Adolphe de Rothschild, Paris, Paris, France